CLINICAL TRIAL: NCT03581942
Title: Phase IB/II Study Combining the PI3K Inhibitor Copanlisib With the BTK Inhibitor Ibrutinib in Patients With Recurrent/Refractory Primary CNS Lymphoma
Brief Title: Copanlisib With Ibrutinib for Patients With Recurrent/ Refractory Primary Central Nervous System Lymphoma (PCNSL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-246
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Refractory/Recurrent Primary Central Nervous System Lymphoma (PCNSL)
Keywords: Copanlisib; Ibrutinib; Recurrent/ Refractory; PCNSL; Brain lymphoma; Primary Central Nervous System Lymphoma; BTK; PI3K
MeSH Terms: interventions — ibrutinib; copanlisib

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase Ib/II trial of the pan-Phosphoinositide 3-kinase (PI3K) inhibitor Copanlisib in combination with the Bruton Tyrosine Kinase (BTK) inhibitor Ibrutinib in patients with recurrent or refractory primary central nervous lymphoma (PCNSL and frail/elderly newly diagnosed PCNSL patients, not eligible to receive standard first-line chemotherapy).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib in combination with Ibrutinib (Experimental): Participants will be assigned to the following dose levels: Dose level 1: Ibrutinib 560 mg daily + Copanlisib 60 mg weekly (3w on/1w off) Dose level 2: Ibrutinib 840 mg daily + Copanlisib 60 mg weekly (3w on/1w off) Dose level -1: Ibrutinib 560 mg daily + Copanlisib 45 mg weekly (3w on/1w off). Phase II: (Simon two-stage design: 14 patients will be treated at the MTD (including 6 patients from the phaseIb portion) If at least 11 patients respond then an additional 19 patients will be accrued to the second stage. Patients in the phase II portion of the trial will receive sequential drug dosing. Patient will be treated in 28-day cycles. During one cycle, only one drug will be administered with a ibrutinib/copanlisib ratio of 1:2. Patients will receive Ibrutinib at 840 mg daily during cycle 1 (day 1 through day 28) (28-day cycles), then copanlisib 60mg weekly on day 1, 8, and 15 during cycle 2 and 3. Patients will then repeat the sequence.
  Interventions: Drug: Ibrutinib; Drug: Copanlisib

INTERVENTIONS:
Drug: Ibrutinib — (MTD) Dose Escalation level 2: Ibrutinib 840 mg daily
Drug: Copanlisib — (MTD) Copanlisib 60 mg weekly (3w on/1w off)

SUMMARY:
The purpose of this study is to test the safety of combined use of the study drugs, copanlisib and ibrutinib, in people with PCNSL.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study must meet ALL the following criteria:

* Men and woman who are at least 18 years of age on the day of consenting to the study.
* Histologically documented PCNSL
* Relapsed/refractory PCNSL or newly diagnosed PCNSL patients who are deemed medically ineligible by the treating investigator (phase II only) to receive standard first-line chemotherapy. All recurrent/refractory patients need to have received at least one prior CNS directed therapy. There is no restriction on the number of recurrences.
* For recurrent/refractory patients, parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI of the brain or head CT) 21 days of study registration. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings consistent with CSF disease 21 days of study registration (at the discretion of the investigator).
* ECOG performance status ≤ 2.
* Life expectancy of > 3 months (in the opinion of the investigator).
* Adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 14 days prior to study registration
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 14 days prior to study registration
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  * Serum creatinine ≤ 2 times the upper limit of normal
  * Creatinine clearance ≥ 30 mL/min
  * Lipase ≤ 1.5 x upper limit of normal
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 30 days (for WOCBP) and 90 days (for men) after the last administration of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

  * The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%), e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence
  * The use of condoms by male patients is required unless the female partner is permanently sterile. Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry
* Must be able to tolerate MRI/CT scans
* Must be able to tolerate lumbar puncture and/or Ommaya taps
* Must have recovered to grade 1 toxicity from prior therapy
* Able to submit up to 20 unstained formalin-fixed, paraffin-embedded (FFPE) slides from the initial or most recent tissue diagnosis for correlative studies

NOTE: Prior autologous stem cell transplant as well as prior radiation to the CNS does NOT prevent patients from enrollment into the trial.

Exclusion Criteria:

Patients eligible for this study must NOT MEET ANY of the following criteria:

* Active concurrent malignancy requiring active therapy
* Newly diagnosed PCNSL who qualify for standard methotrexate-based chemotherapy

Excluded medical conditions:

* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure (New York Heart Association > Class 2), unstable angina, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Uncontrolled hypertension despite optimal medical management (per investigator"s assessment)
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%
* Patient is known to have an uncontrolled active systemic infection (>CTCAE grade 2) and recent infection requiring intravenous anti-infective treatment that was completed ≤14 days before the first dose of study drug
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 3 months before the start of study treatment
* Non-healing wound, ulcer or bone fracture
* Not recovered to a grade 1 from the toxic effects of prior therapy if clinically relevant in the opinion of the investigator (e.g. alopecia)
* Known bleeding diathesis (eg, von Willebrand"s disease) or hemophilia
* Known history of infection with human immunodeficiency virus (HIV) or history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests, or any uncontrolled active systemic infection
* Patient underwent major systemic surgery ≤ 2 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug
* Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction
* Any life-threatening illness, medical condition including uncontrolled diabetes mellitus (DM), uncontrolled hypertension or organ system dysfunction that, in the opinion of the investigator, could compromise the subject"s safety or put the study outcomes at undue risk
* Lactating or pregnant

Excluded previous Therapies and medications:

* Any chemotherapy, external beam radiation therapy, or anticancer antibodies within 21 days of the first dose of study drug
* Prior treatment with a PI3K inhibitor, AKT inhibitor, or mTOR inhibitor (prior ibrutinib exposure is allowed)
* Any targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter
* Use of radio- or toxin-immunoconjugates within 70 days of the first dose of study drug
* Concurrent use of warfarin or other vitamin K antagonists (need to be stopped 7 days prior to starting on trial drug)
* Concurrent use of a strong cytochrome P450 (CYP) 3A4/5 inhibitor and inducers (see Appendix 1) (need to be stopped 2 weeks prior to starting on trial drug)
* Enzyme-inducing antiepileptic drugs (EIAED) need to be discontinued and switched to a nonnon-EIAED 2 weeks prior to starting on trial drug)
* Patient requires more than 4 mg of dexamethasone daily or the equivalent
* Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent. Participants must be off of immunosuppressant therapy for at least 28 days prior to the first dose of the study drug
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration of > 5 mg/day of prednisone) within 28 days of the first dose of study drug
* Prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2026-02-05 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) (phase Ib) | 1 year
  The "3+3" design will be applied in the phase Ib portion of the trial.
overall response rate (ORR) (phase II) | 1 year
  To explore the therapeutic efficacy measured by overall response rate (ORR) of Copanlisib in combination with Ibrutinib in patients with refractory/relapsed PCNSL or newly diagnosed PCNSL not able to tolerate standard chemotherapy (phase II)This study will use the modified International Primary CNS Lymphoma Collaborative Group (IPCG)12.

SECONDARY OUTCOMES:
adverse events in terms of incidence and severity (phase Ib and II) | 2 years
  adverse events at each visit with the NCI CTCAE v4.03 used as a guide for the grading of severity.
progression free survival (PFS) (phase II) | 2 years
  Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause.
duration of response (DOR) (phase II) | 2 years
  Duration of response is defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause.
overall survival (OS) (phase II) | 2 years
  Overall survival time (OS) is defined as the time from treatment start to the date of death due to any cause.
To evaluate cerebral spinal fluid (CSF) pharmacokinetics of Copanlisib and Ibrutinib and correlate with plasma pharmacokinetics (phase Ib) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm